CLINICAL TRIAL: NCT03774680
Title: Polymeric Nanoparticles Loaded With Cetuximab and Decorated With Somatostatin Analogue for Targeting of Colon Cancer
Brief Title: Targeted Polymeric Nanoparticles Loaded With Cetuximab and Decorated With Somatostatin Analogue to Colon Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed A. H. Abdellatif (Other)
Responsible Party: Sponsor-Investigator, Ahmed A. H. Abdellatif, Assistant Professor of Pharmaceutics, Faculty of Pharmacy, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharCetuximab
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Colon Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cetuximab nanoparticles goup (Active Comparator): A group of volunteers infected colon cancer or colorectal cancer received cetuximab in the formulated nanoparticles
  Interventions: Drug: Cetuximab nanoparticles
- Oral approved anticancer drug (Placebo Comparator): A group of volunteers infected with colon cancer or colorectal cancer received placebo anticancer drug.
  Interventions: Drug: Oral approved anticancer drug

INTERVENTIONS:
Drug: Cetuximab nanoparticles — The active group will receive cetuximab in nanoparticles as an anti-microbial drug.
  Other Names: oral capsules
  Arms: Cetuximab nanoparticles goup
Drug: Oral approved anticancer drug — The placebo group will receive topical FDA approved anti-microbial jel in different dosage forms as control drug.
  Other Names: oral capsules
  Arms: Oral approved anticancer drug

SUMMARY:
Due to the great toxicity of chemotherapeutic drugs to both the healthy and cancerous area, the efficient targeting could be of great benefit for a patient with advanced or metastatic tumors. Colorectal cells carry somatostatin receptors which make them a promising target for antitumor therapy since this would reduce side effects and increase drug delivery efficacy to the target site.

DETAILED DESCRIPTION:
The investigator's aim is to deliver polymeric nanoparticles loaded with anti-cancer drug Cetuximab and decorated with somatostatin analogue in the form of oral polymeric nanoparticles, which can release at only above pH 6.8 using ethylcellulose polymer. The polymeric nanoparticles were prepared using the solvent evaporation method, further will be characterized for its drug content, size, encapsulation efficiency and drug-loading using UV spectroscopy. Moreover, the ethylcellulose nanoparticles loaded Cetuximab will release the Cetuximab at pH above 6.8, while can hold the Cetuximab at pH 1.5 which protecting the stomach from the toxicity Cetuximab. Then, the nanoparticles will target the colorectal cancer cells using octreotide, the somatostatin receptor agonist which will lead it to SSTRs overexpressed in colorectal cancer cells. The strategy of deposition of ligand will depend on using the advantage of the positive charge surface of nanoparticles which can absorb the negative charges of the targeting ligands. Final outcomes: this project will present a novel formulation for the treatment of colorectal cancer which can be delivered safely to the patients in a high dose to the affected tumor cells with reduced side effects on the other healthy cells.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colon cancer
* Follow up and collect data for a local and systemic activity of cetuximab
* The systemic oral capsule of cetuximab be also given to enhance the activity as an anti-cancer activities

Exclusion Criteria:

* Peptic ulcer
* Stomach disease
* Colon cancer

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-01-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of pharmacokinetics parameters of Cetuximab for targeted colon cancer | one year
  Determine the bioavailability of Cetuximab after oral and intravenous administration. by measuring the peak levels of Cetuximab after 0.5 to 1.5 hours following ingestion.
  Determine the therapeutic window for Cetuximab after and before formulation in nanoparticles. Determine the different Cetuximab doses, peak plasma levels of Cetuximab for each formula.

CONTACTS AND LOCATIONS:
Locations (4):
- Assiut Clinic, Asyut, Egypt
- Saudi Arabia (3):
  - Buraidah Clinic, Buraidah, Al Qassim
  - Faculty of Pharmacy, Buraidah, Al-Qassim Region
  - Pharmaceutics dept., Faculty of Pharmacy, Qassim University, Buraidah, Al-Qassim Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hafez Abdellatif AA, Abdelhafez WA, Sarhan HA. Somatostatin Decorated Quantum Dots for Targeting of Somatostatin Receptors. Iran J Pharm Res. 2018 Spring;17(2):513-524. PMID 29881409
- [Result] Abdellatif AA, Zayed G, El-Bakry A, Zaky A, Saleem IY, Tawfeek HM. Novel gold nanoparticles coated with somatostatin as a potential delivery system for targeting somatostatin receptors. Drug Dev Ind Pharm. 2016 Nov;42(11):1782-91. doi: 10.3109/03639045.2016.1173052. Epub 2016 May 5. PMID 27032509
- [Result] Allemani C, Weir HK, Carreira H, Harewood R, Spika D, Wang XS, Bannon F, Ahn JV, Johnson CJ, Bonaventure A, Marcos-Gragera R, Stiller C, Azevedo e Silva G, Chen WQ, Ogunbiyi OJ, Rachet B, Soeberg MJ, You H, Matsuda T, Bielska-Lasota M, Storm H, Tucker TC, Coleman MP; CONCORD Working Group. Global surveillance of cancer survival 1995-2009: analysis of individual data for 25,676,887 patients from 279 population-based registries in 67 countries (CONCORD-2). Lancet. 2015 Mar 14;385(9972):977-1010. doi: 10.1016/S0140-6736(14)62038-9. Epub 2014 Nov 26. PMID 25467588